CLINICAL TRIAL: NCT06670742
Title: Gut-muscle Axis: Exploring the Gut Microbiota Influences Host Energy Sources and Exercise Performance Via Modulation of Lactate Metabolism and Utilization
Brief Title: Gut-muscle Axis: Exploring the Gut Microbiota Influences Host Energy Sources and Exercise Performance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Yi-Ju Hsu, Associate Professor, National Taiwan Sport University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NTSUIRB - 112 - 007
Record Dates: First submitted 2024-10-26; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Marathon Runner

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Marathon running group (Experimental): Run 10 kilometers on a treadmill.
  Interventions: Device: running
- General healthy adult group (No Intervention): No intervention will be conducted.

INTERVENTIONS:
Device: running — Running 10 kilometers on a treadmill
  Arms: Marathon running group

SUMMARY:
Through training, the investigators can adjust the composition and functions of gut microbiota. Exercise also alters the body's energy metabolism pathways, which, in turn, impacts the gut microbiota and its metabolic products. Understanding how the body utilizes and regulates energy during exercise is essential for enhancing athletic performance. This study aims to explore the relationships among post-exercise energy metabolites, gut microbiota, and their metabolic products, applying omics technologies in the field of sports science.

This interdisciplinary research will contribute to fields such as exercise physiology, sports nutrition, exercise biochemistry, and sports medicine, providing innovative and practical research insights for advancing sports science in our country.

DETAILED DESCRIPTION:
The gut microbiota, which is comprised of trillions of microbes, is the collective term for the gut microbiota. It establishes a symbiotic relationship with the host and plays a vital role in maintaining host health. Through training, the investigators can adjust the composition and functions of gut microbiota. Exercise also alters the body's energy metabolism pathways, which, in turn, impacts the gut microbiota and its metabolic products. Understanding how the body utilizes and regulates energy during exercise is essential for enhancing athletic performance. This study aims to explore the relationships among post-exercise energy metabolites, gut microbiota, and their metabolic products, applying omics technologies in the field of sports science.

This interdisciplinary research will contribute to fields such as exercise physiology, sports nutrition, exercise biochemistry, and sports medicine, providing innovative and practical research insights for advancing sports science in our country.

ELIGIBILITY:
Marathon Running Group

Inclusion Criteria:

* Training frequency of at least 3 times per week in the past year, with each session involving at least 1 hour of running.
* Participation in at least 2 marathon events within the past 2 years, with a completion time of under 4 hours and 30 minutes for a full marathon, or under 2 hours and 15 minutes for a half marathon.

Exclusion Criteria:

* Excludes individuals with cardiovascular diseases, hypertension, epilepsy, bronchitis, severe asthma, heart disease, inflammatory bowel disease, bacterial or viral infections, disabilities, or chronic bone diseases.
* Habitual smokers.
* Individuals with highly irregular eating habits or sleep patterns due to shift work or night work.
* History of chronic neuro-muscular injuries or disorders in the past 6 months.
* Individuals who have received antibiotic treatment or taken probiotic supplements in the past 6 months.

General Healthy Adult Group

Inclusion Criteria:

* Generally healthy, untrained individuals.

Exclusion Criteria:

* Excludes individuals with cardiovascular diseases, hypertension, epilepsy, bronchitis, severe asthma, heart disease, inflammatory bowel disease, bacterial or viral infections, disabilities, or chronic bone diseases.
* Habitual smokers.
* Individuals with highly irregular eating habits or sleep patterns due to shift work or night work.
* History of chronic neuro-muscular injuries or disorders in the past 6 months.
* Individuals who have received antibiotic treatment or taken probiotic supplements in the past 6 months.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-08 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of lactate | The testing time points are set as follows: before exercise, at the 5-kilometer mark during exercise, immediately after exercise, and at 5, 15, 30, and 60 minutes post-exercise.
  Measure changes in lactate concentration.
Concentration of creatine kinase | The testing time points are set as follows: before exercise, immediately after exercise, and 60 minutes post-exercise.
  Measure changes in creatine kinase concentration.
Concentration of glucose | The testing time points are set as follows: before exercise, immediately after exercise, and 60 minutes post-exercise.
  Measure changes in glucose concentration.
Concentration of creatinine | The testing time points are set as follows: before exercise, immediately after exercise, and 60 minutes post-exercise.
  Measure changes in creatinine concentration.
Concentration of blood urea nitrogen | The testing time points are set as follows: before exercise, immediately after exercise, and 60 minutes post-exercise.
  Measure changes in blood urea nitrogen concentration.
Concentration of lactate dehydrogenase | The testing time points are set as follows: before exercise, immediately after exercise, and 60 minutes post-exercise.
  Measure changes in lactate dehydrogenase concentration.
Concentration of free fatty acid | The testing time points are set as follows: before exercise, immediately after exercise, and 60 minutes post-exercise.
  Measure changes in free fatty acid concentration.
Concentration of cortisol | The testing time points are set as follows: before exercise, immediately after exercise, and 60 minutes post-exercise.
  Measure changes in cortisol concentration.
ood frequency questionnaire(FFQ) | Before exercise
  The participants' diets were assessed using a semiquantitative food frequency questionnaire(FFQ). The FFQ used in this study was validated in a previous study; the questionnaire exhibited reliability and validity for identifying major nutrients in the diets of Taiwanese vegetarians and omnivores.(Chiu TH et al., 2014) In this study, the nutrient analysis programme used to calculate the results of the FFQ was based on Taiwan's Food Composition Database. To assess the intake frequency of each food item, frequencies ranged from "never" or "<1 time per month" to "more than 2 times per day.
Gut microbiota analysis | The testing time points are set as follows: before exercise, immediately after exercise, and at 24 and 48 hours post-exercise.
  Collect participant stool samples for gut microbiota analysis.
Untargeted metabolome analysis | The testing time points are set as follows: before exercise, immediately after exercise, and at 24 and 48 hours post-exercise.
  Collect participant stool samples for metabolome analysis.Metabolite identification aims to analyze the metabolome composition of biological samples, investigate the regulation of metabolic pathways, and explore biochemical mechanisms.

SECONDARY OUTCOMES:
Body composition | Before exercise
  The investigators used the InBody 570 (In-body, Seoul, South Korea), the bioelectrical impedance analyzer (BIA) to measure body composition. The device can screen frequencies of 1, 5, 50, 260, 500 and 1000 kHz within 60 seconds. After cleaning the palms and soles of the feet, the subject stood vertically on the electrodes of the instrument, holding the sensing handle with both hands and keeping the arms away from the body at a 30° angle, and avoided talking or moving during the measurement. The device measured body weight (kg), BMI (kg/m²), fat mass (%), and lean mass (kg).
Rate of Perceived Exertion(RPE) | The testing time points are set as follows: before exercise, at the 5-kilometer mark during exercise, and immediately after exercise.
  Assess perceived exercise intensity.
Heart rate | The testing time points are set as follows: before exercise, at the 5-kilometer mark during exercise, and immediately after exercise.
  Assess changes in heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ju Hsu, Principal Investigator — Associate Professor